CLINICAL TRIAL: NCT04117022
Title: Diabetic Retinopathy Functional Evaluation Study: Monitoring Carotenoid Vitamins Treatment Using ERG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ZeaVision, LLC (Industry)
Collaborators: Northeastern State University (Other); Western University of Health Sciences (Other); Diopsys, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-094
Record Dates: First submitted 2019-10-01; First posted 2019-10-07 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Diabetes; Diabetic Retinopathy
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: Each site will evaluate 15 diabetics after comprehensive ophthalmic examination and with a confirmed diagnosis at least greater than 5 years without retinopathy or mild-moderate retinopathy..Flicker and chromatic ERG, macular pigment optical density, and ultrawide-field undus photography will be conducted at baseline and after 6-months supplementation with a novel multi-component nutritional supplement (DVS)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- supplemented arm (Experimental): Each subject will receive DVS formula, 2 softgels per day for 6 months.
  Interventions: Dietary Supplement: DVS supplementation

INTERVENTIONS:
Dietary Supplement: DVS supplementation — Oral supplement. Each subject will be given the carotenoid supplement of DVS formula. The DVS formula consists of vitamins C, D3 and E (d-α tocopherol), zinc oxide, eicosapentaenoic acid, docosahexaenoic acid, α-lipoic acid (racemic mixture), coenzyme Q10, mixed tocotrienols/tocopherols, zeaxanthin, lutein, benfotiamine, N-acetyl cysteine, grape seed extract, resveratrol, turmeric root extract, green tea leaf, and Pycnogenol (patented French Maritime Pine Bark extract, sp Pinus pinaster, Horphag Research, Geneva, Switzerland). Supplements bottles will be labelled with a unique identification number for each subject and supplied by ZeaVision, LLC, Chesterfield, Missouri, USA. To assure that the participants do not have any issues with the vitamin supplement and to ensure adequate adherence to schedule of vitamin intake the participants will get regular phone calls from the study investigators (once every two weeks).

SUMMARY:
To evaluate the differences in retinal function as measured by ERG in diabetics with and without retinopathy 2) the ability of the Chromatic Electroretinogram (chERG) to detect changes in global retinal function following treatment with Carotenoid Vitamins supplement in patients with diabetic retinopathy (DR). 3) the ability of the Full Field flicker (ffERG) to detect changes in global retinal function following treatment with Carotenoid Vitamins supplement in patients with diabetic retinopathy (DR).

4) Changes in retinal function as observed by OCT-Angiography, following treatment with Carotenoid Vitamins supplement in patients with diabetic retinopathy (DR).

DETAILED DESCRIPTION:
This prospective, study has cross-sectional analysis of ERG functions in a group of diabetics with and without retinopathy. Both Chromatic ERG and Full field ERG (NOVA, Diopsys, Inc. Pine Brook, NJ) will be utilized in the study. Subsequently individuals with an outside normal limit outcome on at least one ERG test will be invited to be part of the longitudinal study. Individuals with abnormal ERG results will be asked to take the carotenoid vitamin supplement (ZeaVision DVS supplement) and the baseline data will be compared to the values at one, three- and six-month follow-up.

The primary endpoint of a patient's follow-up will be at 6 months. The study will be performed at three sites. Western University of Health Sciences, Harpers Pointe Eye Associates (Externship site College of Optometry, Western University of Health Sciences) and Oklahoma College of Optometry, Northeastern State University, Tahlequah, Oklahoma.

The clinical study plan will be reviewed and approved by Eye Care Center of the Western University of Health Sciences Institutional Review Board (IRB). Harpers Pointe Eye Associates will be covered under an externship site of Western University of Health Sciences.

NSUOCO will apply for a separate IRB review at their own site.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-80 years

  1. History of Diabetes for at least > 5years
  2. No retinopathy, Mild or Moderate Non-Proliferative diabetic retinopathy

     * Diabetes without retinopathy (Appendix A)
     * Mild to moderate NPDR as defined by the American Academy of Ophthalmology7 (Appendix A)

Exclusion Criteria:

* • History of any systemic or ophthalmic condition (other than diabetic retinopathy) capable of affecting vision

  * Presence of Diabetic Macular Edema
  * History of intraocular surgery, including macular or panretinal photocoagulation laser (except uncomplicated cataract or keratorefractive surgery more than 6 months prior to enrollment)
  * History of treatment affecting vision, influencing reaction time and/or drugs indicating severe general diseases (eg. Hydroxychloroquine, tamoxifen, dexamethasone, triamcinolone, fluocinolone, etc.)
  * Spherical refraction outside ±5.0 D or cylinder correction outside ±3.0 D
  * Inability to obtain reliable Chromatic ERG test
  * Pregnant and nursing women
  * Allergy to the supplement or any of its ingredients
  * Any subject that all ERG study tests or the OCT angiography cannot be obtained reliably.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Chromatic ERG (ChERG) Outcome Measurements: B wave and PhNR latency (milliseconds) Full field ERG outcome measurements and Chromatic ERG Outcome Measurements | Change from Baseline to 6 months
  The Chromatic Electroretinogram (chERG) and the full field ERG will be recorded using a commercially available system Diopsys® NOVA (Diopsys, Inc. Pine Brook, New Jersey). The Red-Blue stimulus will be presented using a mini-Ganzfeld handheld device. The entire process consists of two tests per eye, with twenty-five seconds allocated for each test; thus, the total duration of the test is one hundred seconds. The chERG will be consecutively recorded from both eyes by means of proprietary adhesive skin electrodes on the lower eyelid and forehead.
Full-field flicker ERG (ffERG) Measurements: magnitude (microvolts) and the phase (milliseconds) and the area ratio for magnitude and the area ratio for Phase | Change from Baseline to 6 months
  The Flicker ERG will be recorded using a commercially available system, Diopsys® NOVA (Diopsys, Inc., Pine brook, NJ), version 2.19.19778.7332). The Flicker ERG will be consecutively recorded from both eyes by means of adhesive skin electrodes on the lower eyelid and skin. The stimulus will consist of white flashes flickering at 32 Hz over a white background as well as a sequence of 6 steps of increasing luminance.

SECONDARY OUTCOMES:
Macular pigment optical density (MPOD in relative density units) | Change from Baseline to 6 months
  Subjects are asked to identify when they detect a flickering stimulus of varying intensity, allowing determination of relative density of xanthophyll macular pigments.
Optical coherence tomography angiography (OCTA): radial macular and optic nerve capillary density (number/square millimeter) | Change from Baseline to 6 months
  OCT angiography measurements will be performed using the Angiovue OCT by Optovue CA. It is a camera system that utilizes interferometry to measure the thickness and vascular profile of the macula and the optic nerve, allowing measurement of radial capillary count in both macula and the peripapillary optic nerve head region

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Lighthizer, OD, Study Chair — Northeastern State University, School of Optometry; Pinakin Davey, OD, PhD, Principal Investigator — Western University of Health Sciences, College of Optometry
Locations (2):
- United States (2):
  - Western Universit5y of Health Sciences, College of Optometry, Pomona, California
  - Oklahoma College of Optometry, Northeastern State University, Tahlequah, Oklahoma

IPD SHARING:
Plan to Share IPD: No
anonymized data for statistical analysis only

REFERENCES:
- [Result] Chous AP, Richer SP, Gerson JD, Kowluru RA. The Diabetes Visual Function Supplement Study (DiVFuSS). Br J Ophthalmol. 2016 Feb;100(2):227-34. doi: 10.1136/bjophthalmol-2014-306534. Epub 2015 Jun 18. PMID 26089210